CLINICAL TRIAL: NCT03979976
Title: Ramipril Improves Endothelial Function and Endothelial Progenitor Cells in Patients With Systemic Lupus Erythematosus: a Randomized and Controlled Study.
Brief Title: Ramipril, Endothelial Function and Endothelial Progenitor Cells in Patients With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Emilia Inoue Sato, Full professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ramipril.unifesp
Record Dates: First submitted 2013-09-18; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; endothelium; ramipril
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Ramipril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ramipril group (Active Comparator): Use of ramipril 10mg/day per 12 weeks
  Interventions: Drug: Ramipril
- Control Group (No Intervention): Without ramipril

INTERVENTIONS:
Drug: Ramipril — Use of ramipril 10mg/day per 12 weeks. Telephone contact was made in the second and sixth week, to ask about possible side effects and ensure adherence
  Other Names: angiotensin-converting enzyme inhibitor (ACEI)
  Arms: ramipril group

SUMMARY:
The aim of this study was to evaluate the effect of ramipril on the endothelial function and on the number of endothelial progenitor cells (EPCs) in systemic lupus erythematosus (SLE) patients.

DETAILED DESCRIPTION:
The early detection of additional risk factor for cardiovascular diseases (CVD) such as endothelial dysfunction and low number of EPC in SLE patients, and an intervention proven effective could reduce the cardiovascular morbidity and mortality. No study assessed the effect of ramipril on endothelial function and EPCs in SLE patients.

ELIGIBILITY:
Inclusion Criteria:

* SLE according 1997 modified American College Rheumatology criteria
* age older than 18 years
* stable treatment for lupus for at least 3 months

Exclusion Criteria:

* previous coronary artery disease
* hypertension
* dyslipidemia (LDL>149 mg/dL)
* renal insufficiency (creatinine ≥1.4 mg/dL)
* diabetes
* smoking
* obesity (BMI≥30)
* pregnancy
* menopause
* patients taking statins or angiotensin convertor enzyme inhibitor within the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Endothelial function - Variation of Flow mediated dilation percentage | 12 weeks
  Patients were evaluated at baseline and after 12 weeks by high-resolution ultrasound of brachial artery in resting conditions, after reactive hyperaemia (flow-mediated dilation-FMD) and after oral glyceryl trinitrate to assess endothelial function
Number of endothelial progenitor cells (EPC) | 12 weeks
  Patients were evaluated at baseline and after 12 weeks. EPCs were evaluated by flow cytometry using anti-CD34 (cluster of differentiation 34) (FITC), anti-CD133 (PE) and anti-kinase domain receptor (KDR) (APC) and by cell culture with quantification of colony formation units (CFUs).

CONTACTS AND LOCATIONS:
Overall Officials: Emilia I Sato, MD, PhD, Study Chair — Universidade Federal de São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliveira ACD, Arismendi MI, Machado LSG, Sato EI. Ramipril Improves Endothelial Function and Increases the Number of Endothelial Progenitor Cells in Patients With Systemic Lupus Erythematosus. J Clin Rheumatol. 2022 Oct 1;28(7):349-353. doi: 10.1097/RHU.0000000000001869. Epub 2022 Jun 8. PMID 35662232